CLINICAL TRIAL: NCT06113549
Title: Grip on Knee Osteoarthritis; DIstraction Versus Arthroplasty (GODIVA) for Young Knee Osteoarthritis Patients in Regular Care
Brief Title: Grip on Knee Osteoarthritis; DIstraction Versus Arthroplasty
Acronym: GODIVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Paco M.J. Welsing, Associate Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-732/G
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; knee prosthesis indication
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Knee Prosthesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee Joint Distraction (KD) (Experimental): Knee joint distraction (KJD) is a joint-preserving treatment for knee OA for younger patients, where the knee joint is temporarily fully unloaded by distraction of tibia and femur, using an external fixation frame. KJD treatment is performed according to the current approved concept NOV recommendations for clinical practice.
  Interventions: Procedure: Knee Joint Distraction (KD)
- Knee Prosthesis (Active Comparator): KP is indicated and surgically implanted according to regular clinical practice (can be a total- or unicompartmental KP, in line with local practice in consultation with the patient and conform the national guideline by Dutch orthopaedic society (NOV)).
  Interventions: Procedure: Knee Prosthesis

INTERVENTIONS:
Procedure: Knee Joint Distraction (KD) — Knee joint distraction (KJD) is a joint-preserving treatment for knee OA for younger patients, where the knee joint is temporarily fully unloaded by distraction of tibia and femur, using an external fixation frame.KJD treatment is performed according to the current approved concept NOV recommendations for clinical practice.
  Arms: Knee Joint Distraction (KD)
Procedure: Knee Prosthesis — A total or unicompartmental knee prosthesis
  Arms: Knee Prosthesis

SUMMARY:
The goal of this pragmatic, open, (1:1) randomized, multi-centre, non-inferiority trial is to to determine whether knee-joint distraction (KD) is non-inferior on patient reported effectiveness as compared to a knee-prosthesis (KP; i.e. usual care) for relatively young patients with end-stage knee Osteoarthritis (OA).

The main question[s] it aims to answer are:

* Is KD non-inferior to KP regarding pain, function and stiffness (as indicated by the total score on the total Western Ontario and McMaster Universities Osteoarthritis Index' (WOMAC), with a non-inferiority limit of 15 points) at 2 years?
* Is KD non-inferior to KP regarding Quality of Life (36-Item Short Form Health Survey, (SF36), Physical- and Mental- Component Summary (PCS/MCS), with a non-inferiority limit of 10 points) at 2 years?
* Does KD lead to regeneration of tissue (increase in minimum joint-space-width > 0.05mm on x-ray) over 2 years?

Participants will be allocated to undergo either a knee joint distraction or prosthesis (total- or unicompartmental KP according to orthopedic surgeon/patients discretion), and groups will be compared using will be compared between groups using (multivariable) random effects (mixed) modelling to account for the nested and longitudinal structure of the data over the 24 months follow-up. The stratification factors for randomization, center (using a random intercept) and gender, as well as a limited number of a priori defined prognostic factors (i.e. baseline WOMAC total score, age, BMI, severity of cartilage damage) will be accounted for in this analysis. The difference in mean total WOMAC score at 24 months between treatment groups will be estimated from this model with a 95% confidence interval (CI) and non-inferiority will be determined using the lower limit of this confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee OA
* Age ≤ 65 years and ≥ 18 years
* Persistent, refractory pain, insufficiently responding to conservative or previous surgical therapy
* Structural OA joint damage, indicated by a K&L grade of at least 2 as determined by the orthopedic surgeon in line with NOV recommendations.
* Able to wear an external fixator and care for it for 6 weeks
* Accepting that the maximal effect of KJD is not present directly after removal of the frame but may take months after frame removal
* Sufficient joint stability (according to the orthopedic surgeon's judgement)
* Flexion (>100 degrees) and extension range (<10 degrees)
* Weight and BMI <120 kg and <35 kg/m2, respectively
* Sufficient understanding of the Dutch language
* Signed informed consent

Exclusion criteria:

* Surgical intervention in last 6 months
* Leg-axis deviation > 10 degrees (as determined by the orthopedic surgeon)
* Serious osteopenia making placing bone-pins and wearing a frame into a risk (according to the orthopedic surgeon's judgement)
* Coagulation problems making occurrence of thrombosis or embolies into a risk (according to the orthopedic surgeon's judgement)
* Existing endoprosthesis at any other joint (e.g. hip or contralateral knee) to prevent infection of existing prosthesis
* History or presence of joint infection/inflammation
* Hypersensitivity to antibiotics
* Presence of systemic inflammatory disease, like rheumatoid arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
WOMAC total Score | at 24 months
  Western Ontario and McMaster Universities Osteoarthritis Index' (WOMAC) total score (scale 0-100, higher scores indicate improvement), with a non-inferiority limit of 15 points

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQol) | 24 months
  SF36 physical component score and mental component score (0-100)

DOCUMENTS (1):
  • Study Protocol (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT06113549/Prot_000.pdf